CLINICAL TRIAL: NCT04111354
Title: Early Mobilization After Pacemaker Implantation.
Acronym: EMAPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jiri Smid, M.D., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Early mobilization 14-3-2019
Record Dates: First submitted 2019-09-06; First posted 2019-10-01 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pacemaker Complication; Mobilization
Keywords: pacemaker; implantation; mobilization; complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-term (4-hours) immobilization. (Active Comparator): Short-term (4-hours) immobilization after primary pacemaker implantation.
  Interventions: Device: Pacemaker implantation
- Long-term (16-24 hours) immobilization. (Active Comparator): Long-term (16-24 hours) immobilization after primary pacemaker implantation.
  Interventions: Device: Pacemaker implantation

INTERVENTIONS:
Device: Pacemaker implantation — Pacemaker implantation

SUMMARY:
Permanent pacemaker implantation is one of the most common arrhythmological procedure. This procedure is usually accompanied by a minimum of 2-3 days hospitalization, with immobilization of patients (supine) for 16-24 hours. The optimal duration of patient´s immobilization is not determined. There is also no recommendation from individual manufacturers of pacemakers for the duration of immobilization after pacemaker implantation. The length of immobilization is based rather on the tradition established at the time of using electrodes with passive fixation. The aim of our prospective, randomized study (EMAPI) is to compare the safety of short-term (4-hours) immobilization with long-term (16-24 hours) immobilization after primary pacemaker implantation. Septal position will be used for right ventricular electrode.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older.
2. Indication for permanent pacemaker implantation.
3. Mobile and compliant patient.
4. Willing and able to give written informed consent.

Exclusion Criteria:

1. Imobile and noncompliant patient.
2. Indication of CRT implantation.
3. Upgrade or revision of implanted devise.
4. Contraindications to pacemaker implantation.
5. Gravidity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of incidence of adverse events from secondary outcomes depending on the length of immobilization (early vs. late). | 6 months
  Comparsion of incidence of dislodgement of atrial electrode, dislodgement of ventricular electrode in septal position, hematoma surgically treated or requiring blood transfusions, pneumothorax, pocket infection, others complications

SECONDARY OUTCOMES:
Incidence of atrial lead dislodgement. | 6 months
  comparsion of early vs. late mobilization
Incidence of ventricular lead dislodgement. | 6 months
  comparsion of early vs. late mobilization
Incidence of hematoma (surgically treated or requiring blood transfusions.) | 6 months
  comparsion of early vs. late mobilization
Incidence of pneumothorax. | 24 hours
  comparsion of early vs. late mobilization
Incidence of pocket infection. | 6 months
  comparsion of early vs. late mobilization
Incidence of others complications. | 6 months
  comparsion of early vs. late mobilization, (mechanical, extracardiac complication etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Jiri Smid, Cardiology department, University Hospital and Faculty of Medicine in Pilsen, Charles University, Czech Republic, Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: No